CLINICAL TRIAL: NCT04038073
Title: Toll-Like Receptor Polymorphism, Antinuclear Antibodies and Beta-hemolytic Group A Streptococcus Infections in Attention-Deficit/Hyperactivity Disorder: an Observational Study
Brief Title: TLR Polymorphism, ASO and Beta-hemolytic Group A Streptococcus Infections in ADHD: an Observational Study
Acronym: TLR;
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Francesco Oliva, Research Assistant Professor, University of Turin, Italy
Other Study IDs: ADHD_TLR
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Attention Deficit-Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADHD: Attention Deficit/Hyperactivity Disorder
  Interventions: Diagnostic Test: Antistreptolysin O Test; Diagnostic Test: Anti-Deoxyribonuclease B; Diagnostic Test: TLR, MyD88, IRAK-4 polymorphism; Diagnostic Test: Anti-Basal Ganglia Antibody

INTERVENTIONS:
Diagnostic Test: Antistreptolysin O Test — Test to evaluate of any histories of streptococcal infections
  Other Names: ASO
Diagnostic Test: Anti-Deoxyribonuclease B — Test to evaluate of any histories of streptococcal infections
  Other Names: Anti-DNase B
Diagnostic Test: TLR, MyD88, IRAK-4 polymorphism — Test to evaluate of the frequency and types of genetic alterations of innate immunity
Diagnostic Test: Anti-Basal Ganglia Antibody — Test to evaluate the autoimmune component
  Other Names: ABGA

SUMMARY:
The aim of this observational cross-sectional study is to evaluate the streptococcal infection (clinical history, ASLO title and anti-DNAse title B) and autoimmunity (ABGA antibodies) in a sample of 100 adult patients diagnosed with ADHD (ie in patients in whom the disorder is permanent). Another objective will be to evaluate the frequency and types of genetic alterations of innate immunity (TLR polymorphisms, MyD88, IRAK-4) that can determine an infantile susceptibility to gram positive infections (ie S. pyogenes, S. pneumoniae, S. aureus) and the possible relationship between these elements, also in relation to comorbidity with other ABGA-related pathologies, to identify a possible pathogenetic immune mechanism of ADHD. Prevalence data will be obtained on an outpatient ADHD population for previous (history) and recent streptococcal infection (ASLO and Anti-DNAsiB), for the detection of ABGA and for the co-presence of other ABGA-related pathologies. By comparing the subgroups obtained by dividing the results on the basis of the positive infectious history, anti-streptococcus, autoantibody and comorbidity titers, it will be possible to assess whether the elevation of the ABGA titer is only linked to the previous/current infection ("infectious" group) or if there is a subpopulation of ADHD patients presenting pathological elevation of ABGA titers in the absence of infectious pictures ("immune" group). Furthermore, it is expected that the comparison of the descriptive polymorphisms TLR, MyD88 and IRAK-4 between the "infectious" and "immune" group may show a predisposition in subjects of the "immune" group.

DETAILED DESCRIPTION:
Attention Deficit / Hyperactivity Disorder (ADHD) is the most widespread neurodevelopmental disorder (prevalence 3-7% in preschool age) and is characterized by persistent inattention and / or hyperactivity-impulsivity which results in significant impairment in at least two areas of operation (usually scholastic / working and relational) with consequent impact even on the child's self-esteem. It is estimated that one-third of children with ADHD continue to be affected in adulthood and that around one-third have remission of symptoms with persisting changes in functioning and development of psychiatric disorders in adulthood (eg anxiety disorders mood and personality). The pathogenetic model of ADHD is still poorly characterized: several biological, psychological and environmental causes have been identified that would seem to interact in a complex way in determining the pathology. Several studies have hypothesized and confirmed an association between streptococcal infections, increased titer of antibodies to the basal nuclei (ABGA), different neurological and psychiatric disorders (eg, Sydenham chorea, Tic Disorders, Obsessive-Compulsive Disorder) and ADHD. ADHD is diagnosed in 40% of autoimmune neuropsychiatric disorders associated with streptococcal infection (PANDAS) and Sydenham Korea and a temporal connection between onset / exacerbation of ADHD and pharyngeal streptococcal infection has been described in literature. High titers of anti-streptococcal antibodies and larger size of putamen and pallidum were found in ADHD patients. However, the permanence of symptoms ADHD at a distance from streptococcal infection has led to hypothesize, as already done for PANDAS and Sydenham Korea, a miminking mechanism with consequent cross-reactivity towards host tissues that would support an autoimmune disorder characterized by the production of ABGA.

According to some authors, therefore, ADHD and other ABGA-related neurological and psychiatric disorders (eg, Sydenham Korea, Tic Disorders, Obsessive-Compulsive Disorder) would be different phenotypic manifestations of a common immunological disorder affecting the nuclei of the base, triggered from group A beta-hemolytic streptococcus. The search for ABGA in ADHD patients with Tic Disorders and Obsessive-Compulsive Disorder has largely confirmed this hypothesis, however, the finding of ABGA titres in ADHD patients without comorbidities with other ABGA-related disorders is still controversial. A first study found no differences significant in terms of ABGA positivity frequency among ADHD patients without ABGA related disorders and controls while a more recent study conducted confirmed that children with ADHD without ABGA-related disorders are more frequently positive for ABGA than the control group (30% vs 4.8%; χ2 = 4.33; p = 0.04) and that, among these, those with Anti-Streptolysinic Title (ASLO) show significantly higher percentages of ABGA positivity (χ2 = 10.95; p <.001). On the other hand, greater susceptibility by ADHD patients to contracting streptococcal infections was confirmed by the finding of significantly higher titers of ASLO and anti-DNAse B in ADHD patients.

The predisposition to infections and the high familiarity of ADHD (90% of cases have at least one affected parent), suggest an immune pathogenetic mechanism based on a genetic predisposition.

Although several studies have established, in an inconclusive way, a relationship between ADHD and some regulatory genes, the major histocompatibility complex (MHC), such as HLA-DR4, HLA-DRB1 and C4B, to date no one has yet evaluated the role of Toll-type receptor (TLR) genes, which are more responsible for innate immunity, ie the recognition of pathogenic structural molecules. In particular, some variants of the TLR genes could affect the immune response to strepotococcus or other pathogens, favoring damage to the nuclei of the base which would in turn lead to ADHD symptoms. Recently, an association between susceptibility to serious or recurrent infections from group A beta-hemolytic streptococcus, Streptococcus pneumoniae, Haemophilus influenza and particular polymorphisms of TLR2, TLR4 and TLR9 has been demonstrated. The altered functioning consequent to these TLR polymorphisms could explain both the vulnerability to certain types of pathogens responsible for lesions to the central nervous system (among which the most studied so far is Group A beta-hemolytic streptococcus), whether the incongruous or excessive immune activation even in the absence of contact with pathogens producing autoantibodies against the nerve structures of the base nuclei.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ADHD according to DSM-5 criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with ADHD disgnosis (according to DSM-5 criteria) will be recruited for a single blood sample.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Antistreptolysin O and Anti-Deoxyribonuclease B | up to 1 year till the end of the study
  diagnostic blood sample test to measure streptococcal infections
Measurement of TLR, MyD88, IRAK-4 polymorphism | up to 1 year till the end of the study
  diagnostic blood sample test to measure genetic alterations of innate immunity
Measurement of Anti-Basal Ganglia Antibody | up to 1 year till the end of the study
  diagnostic blood sample test to assess the autoimmune component

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Oliva, Principal Investigator — University of Turin, Italy
Locations (1):
- AOU San Luigi Gonzaga di Orbassano, Orbassano, Torino, Italy

IPD SHARING:
Plan to Share IPD: No